CLINICAL TRIAL: NCT04558138
Title: A Randomized Controlled Trial in Patients Undergoing Immediate Implant-Based Breast Reconstruction Utilizing an Enhanced Recovery Pathway Comparing Outcomes and Patient Satisfaction Based on Time of Discharge
Brief Title: RCT Implant Based Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-1055.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-08-17; First posted 2020-09-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Mastectomy
Keywords: Reconstruction

STUDY DESIGN:
Intervention Model Description: After consent, patients will be randomized into one of two groups, either discharged day of surgery, or discharged day after surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discharge day of surgery (Experimental): Patient discharges day of surgery and given surveys to complete at home on post operative day (POD) #1 and #7.
  Interventions: Other: Discharge timing
- Discharge post operative day 1 (No Intervention): Patient Discharges POD #1 and completes survey prior to discharge. Patient given surveys to complete POD #7 at home.

INTERVENTIONS:
Other: Discharge timing — Patients will be discharged home on the day of surgery as opposed to POD #1
  Arms: Discharge day of surgery

SUMMARY:
The main objective of this study is to evaluate patients undergoing mastectomy with immediate implant-based breast reconstruction and compare the outcomes of patients who are discharged the day of surgery versus patients who are discharged on post-operative day one. The primary aim of the study will be to compare the postoperative outcomes and complications between the two study groups within 30 days of discharge. The secondary aims of the study will be to compare patient satisfaction, quality of life and discharge perceptions.

DETAILED DESCRIPTION:
Traditionally patients undergoing mastectomy with immediate implant-based breast reconstruction were admitted to the hospital overnight. However, recent retrospective studies utilizing ERAS protocols have reported same day discharge as a possibility for this patient population. ERAS protocols for breast cancer surgery and reconstruction are becoming more popular. This along with the increasing utilization of prepectoral breast reconstruction that is associated with less postoperative pain and opioid use, are promising avenues to decrease the need for overnight hospital stay. If it can be shown that discharge on the same day of surgery does not pose any major risks compared to discharge on post-operative day one, there is the potential to decrease length of hospital stay, improve hospital capacity and dramatically decrease costs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo immediate, (unilateral or bilateral)implant-based breast reconstruction following mastectomy for breast cancer or prophylaxis at the University of Colorado Anschutz Medical Campus and Highlands Ranch Campus.
2. Patients undergoing sub-pectoral and pre-pectoral breast implant reconstructive techniques will be both included.
3. All adult (>18 years old), female patients who will undergo mastectomy for breast cancer or prophylaxis and immediate implant-based reconstruction who are able to complete surveys independently will be eligible for the study.
4. English and Spanish speaking
5. Patients will be included regardless of their current chemoradiation plan

Exclusion Criteria:

1. Age > 80 years
2. ASA 4
3. suboxone use
4. documented substance use disorder as defined by the DSM-5 (I.e. alcohol use disorder, opioid use disodrer, cocaine use disorder, etc). Marijuana use will not be considered a substance use disorder
5. OSA requiring CPAP
6. recent pneumonia (within 6 weeks)
7. BMI > 45 kg/m2 with any co-morbid condition that is not well controlled
8. poorly controlled diabetes (HgbA1c > 9)
9. Not English or Spanish speaking

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Rate of post-operative complications surgical site infection | Up to 30 Days
  Assessed by patient report
Number of Participants with Post-operative hematoma | Up to 30 Days
  Assessed by patient report
Number of Participants with Post-operative blood clots | Up to 30 Days
  Assessed by patient report
Number of Participants with Post-operative emergency department visits | Up to 30 Days
  Assessed by patient report
Number of Participants with Post-operative hospital readmissions | Up to 30 Days
  Assessed by patient report
Number of Participants with Post-operative re-operation | Up to 30 Days
  Assessed by patient report

SECONDARY OUTCOMES:
Pain Score | Up to 30 Days
  Pain control, as measured by a visual analog Numeric Pain Scale (NPS) number ranging from 0 (no pain at all) to 10 (worst pain ever) between the two groups.
Opioid Consumption | Post-Operative day 7
  The following information will be collected from a combination of patient reported information and electronic medical review: amount of supplemental postoperative opioid analgesia (both intravenous and oral) used by the study participant from postoperative days 0 to 7.
Opioid adverse effects | Up to 30 Days
  The following effects/symptoms will be recorded as YES or NO if required admission to the hospital for management including use of IV medications: nausea, vomiting, constipation and urinary retention.
Quality of life perceptions: QoR-15 | Up to 30 Days
  QoR-15: This scale will be utilized to evaluate patient satisfaction. It captures patient reported postoperative assessment of various dimensions of health including patient support, comfort, emotions, physical independence, and pain. Patients rate each of the 15 statements from 1 (never) to 10 (always).
Discharge perceptions | Post-Operative day 7
  Group A: Discharged the same day of surgery will be asked the following questions on postoperative 7:
  Did you feel that you were discharge home at the appropriate time?
  How uncomfortable were you the night of surgery, as measured by a visual analog NPS number ranging from 0 (not uncomfortable) to 10 (extremely uncomfortable)?
  What was the main benefit of going home right after surgery?
  What was your biggest complaint about being at home right after surgery?
  Group B: Patients admitted after surgery will be asked the following questions on postoperative 7:
  Did you feel that you were discharge home at the appropriate time?
  How uncomfortable were you the night of surgery, as measured by a visual analog NPS number ranging from 0 (not uncomfortable) to 10 (extremely uncomfortable)?
  What was the main benefit of being admitted to the hospital after surgery?
  What was your biggest complaint about being at the hospital after surgery?
Quality of life perceptions: PROMIS-29 | Up to 30 Days
  PROMIS-29: A generic health-related quality of life survey, assesses each of the 7 PROMIS domains with 4 questions. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity part of the PROMIS-29 (with 0 being "no pain" and 10 being "worst imaginable pain")

CONTACTS AND LOCATIONS:
Overall Officials: Christodoulos Kaotzanis, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No